CLINICAL TRIAL: NCT02340117
Title: Phase II Study of Combined Targeted p53 Gene Therapy (SGT-53) Plus Gemcitabine/Nab-Paclitaxel for Treatment of Metastatic Pancreatic Cancer
Brief Title: Study of Combined SGT-53 Plus Gemcitabine/Nab-Paclitaxel for Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT53-02-1
Record Dates: First submitted 2014-12-18; First posted 2015-01-16 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGT-53 with gemcitabine/nab-paclitaxel (Experimental): A course of therapy will include 7 weeks of treatment. SGT-53, at 3.6 mg DNA/infusion, will be administered bi-weekly on days 1 and 5 in weeks 1-3, weekly on day 3 in week 4, and weekly on day 1 in weeks 5-7. Patients who are responding to treatment may receive two additional courses (7 weeks) of SGT-53/gemcitabine/nab-paclitaxel therapy at investigator discretion. If still responding to treatment, they may continue on SGT-53/gemcitabine/nab-paclitaxel at investigator discretion with the approval of the sponsor.
  Interventions: Genetic: SGT-53; Drug: nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Genetic: SGT-53 — The dose of SGT-53 will be 3.6 mg DNA/infusion. If necessary, the dose of SGT-53 can be de-escalated to 2.4 mg, 1.2 mg or 0.6 mg DNA per infusion in the event that increased toxicity probably or definitely related to SGT-53 is observed with the combination.
Drug: nab-paclitaxel — The dose of nab-paclitaxel will be 125 mg/m² and will be administered once weekly (day 3) in weeks 1, 2, 3, 5, 6 and 7. If increased toxicities related to administration of nab-paclitaxel is observed, the dose of nab-paclitaxel can be reduced to 100 or 75 mg/m² when appropriate.
  Other Names: Abraxane ABI-007; Albumin-bound paclitaxel
Drug: Gemcitabine — The dose of gemcitabine will be 1000 mg/m² and will be administered once weekly (day 3) in weeks 1, 2, 3, 5, 6 and 7, after the administration of nab-paclitaxel. If increased toxicities related to administration of gemcitabine is observed, the dose of gemcitabine can be reduced to 800 or 600 mg/m² when appropriate.
  Other Names: Gemzar

SUMMARY:
This clinical trial is an open label Phase II study of the combination of intravenously administered SGT-53 and gemcitabine/nab-paclitaxel in patients with metastatic pancreatic cancer. The objective of the study is to evaluate the safety, tolerability, toxicity and efficacy (specifically Progression Free Survival at 5.5 month (PFS5.5mos)) of this combination therapy.

DETAILED DESCRIPTION:
The p53 is a vital human tumor suppressor gene. Loss of p53 suppressor function is present in the majority of human cancers. The p53 protein has a diverse range of functions including regulation of cell cycle checkpoints, cell death (apoptosis), senescence, DNA repair, maintenance of genomic integrity, and control of angiogenesis. Abnormalities of the p53 gene may impact the efficacy of standard anticancer treatments such as radiation and chemotherapy. P53 mutation and pathway dysfunction are associated with poor clinical outcomes and the presence of the p53 mutation correlates with resistance to chemotherapy and radiation. The development of somatic gene therapy has created the potential to restore wild type function of p53. SGT-53 is a complex of cationic liposome encapsulating a normal human wild type p53 DNA sequence in a plasmid backbone. This complex has been shown to efficiently and specifically deliver the p53 cDNA to the tumor cells. Introduction of the p53 cDNA sequence is expected to restore wtp53 function in the apoptotic pathway. P53 restoration has been shown most effective in enhancing cytotoxicity in combination with an agent which results in DNA damage or initiates apoptosis. This is a Phase II clinical trial of SGT-53 plus the recently approved chemotherapeutic combination of gemcitabine/Abraxane® (nab-paclitaxel) in patients with confirmed metastatic pancreatic cancer. In addition to determining Progression Free Survival at 5.5 months (PFS5.5mos), this trial will evaluate the response rate, overall survival and time to progression as well as the tolerability and safety of SGT-53 in combination with gemcitabine/nab-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic diagnosis of stage IV metastatic pancreatic adenocarcinoma.
* One or more tumors measurable on CT scan.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Life expectancy of at least 3 months.
* Age ≥ 18 years.
* Signed, written IRB-approved informed consent.
* A negative pregnancy test (if female and of child-bearing potential).
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times upper limit of normal
  * AST (SGOT), ALT (SGPT) ≤ 3.0 x ULN
  * Serum creatinine ≤ 1.5 X ULN
* Acceptable hematologic status:

  * Absolute neutrophil count ≥ 1500 cells/mm³
  * Platelet count ≥ 100,000 (plt/mm³)
  * Hemoglobin ≥ 10 g/dL
* Acceptable blood sugar control

  *Fasting glucose value ≤ 160 mg/dL
* Urinalysis: No clinically significant abnormalities.
* PT and PTT ≤ 1.5 X ULN
* For men and women of child-producing potential, willingness to use of effective contraceptive methods during the study.
* NOT have received any prior cytotoxic chemotherapy or investigational therapy. However, this study may be used as 2nd line treatment of patients who progressed on or were intolerant of 1st line FOLFIRINOX for the primary or metastatic disease. Prior treatment with gemcitabine administered as radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* They also must NOT have received chemotherapy, radiotherapy, surgery or investigational therapy for the treatment of metastatic disease.
* Organ function characterized by ≤ Grade 1.

Exclusion Criteria:

* Patient has received any prior cytotoxic chemotherapy for pancreatic cancer with the exception of patients who progressed on or were intolerant of 1st line FOLFIRINOX in primary or metastatic disease. Prior treatment with gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. Patients who previously had and were treated with standard therapy for non-pancreatic cancer will be evaluated for entry into the trial on a case-by-case basis.
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, unstable angina (chest pain greater than three times weekly while on therapy), evidence of ischemia on ECG, or abnormal stress echocardiogram with evidence of ischemia, or LVEF < 50%.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Treated with antibiotics for infection within one week prior to study entry.
* Fever (> 38.1°C)
* Have hematological malignancy
* Have diastolic blood pressure of > 90 mm Hg resting at baseline despite medication.
* Pregnant or nursing women.
* Treatment with surgery, or investigational therapy within 28 days prior to study entry or radiation therapy within 6 months prior to study entry.
* Have received chemotherapy, radiotherapy, surgery or investigational therapy for the treatment of metastatic disease.
* Unwillingness or inability to comply with procedures required in this protocol.
* Known infection with HIV, Hepatitis B, or Hepatitis C.
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* Patients who are currently receiving any other investigational agent.
* Patients who are currently taking Coumadin or Coumadin derivatives other than to maintain patency of venous access lines.
* Receiving systemic steroids or other chronic immunosuppressive medications within 30 days prior to study entry
* Receiving hematopoietic growth factors on a regular basis
* Had within six months prior to enrollment any of the following:

  * Cerebrovascular accident
  * Uncontrolled congestive heart failure
* Have significant baseline neuropathies
* Requires renal dialysis
* Had prior exposure to gene vector delivery products
* Had previously experienced a severe hypersensitivity reaction to gemcitabine or nab-paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 5.5 months | 5.5 months
  PFS5.5mos will be assessed by objective radiographic assessment
Objective response rate (ORR) | Up to 5 years
  ORR will be assessed by objective radiographic assessment using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 5 years
  Progression free survival (PFS) will be defined as the time from registration until confirmed tumor progression or death, whichever occurs first.
Overall survival (OS) | Up to 5 years
  Survival will be defined as the time from the date of registration to the date of death (any cause).
Time to disease progression (TTP) | Up to 5 years
  Time to disease progression is defined as the time from registration until confirmed tumor progression, but not including deaths.
Disease control rate (DCR) | 16 weeks
  Disease control rate (SD for ≥16 weeks plus CR and PR) will be analyzed using Kaplan-Meier methods.
Duration of disease control | Up to 5 years
  Disease control duration is measured from the time of registration until documented confirmed tumor progression.
Adverse events | Study drug initiation through 30 days after the last dose of study drug or end of treatment, whichever is later.
  Safety will be evaluated by the incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs), physical examination, laboratory abnormalities during study drug dosing and percentage of patients experiencing dose modifications, interruptions, and/or discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Center
Locations (1):
- Mary Crowley Cancer Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided